CLINICAL TRIAL: NCT04541472
Title: Influence of the COVId-19 Pandemic on the STRESS of Dental Surgeons
Brief Title: Influence of the COVId-19 Pandemic on the STRESS of Dental Surgeons (COVISTRESS - Dental Surgery)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2020 COVISTRESS Dental Surgery
Record Dates: First submitted 2020-09-07; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Dental Surgeon
Keywords: COVID-19; Dental surgery; Stress
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus has caused containment of more than half of the world's population and a major and rapid reorganization of clinical and support services. The spread of coronavirus (COVID-19) has posed significant challenges for dental surgeons and associates who are at high risk of COVID-19 infection due to close face-to-face contact. However, there is currently no data on the influence of this epidemic on the practice and feelings of dental surgeons and associates

DETAILED DESCRIPTION:
This is an observational study by REDCap questionnaire® via an internet link, which will be distributed to dental surgeons and associates by any means The self-survey will assess stress, working conditions and changes in practices related to the coronavirus outbreak. This Dental Surgery questionnaire includes 16 questions

ELIGIBILITY:
Inclusion Criteria:

* All dental surgeons and associates volunteers to participate

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Dental surgeons and associates
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Stress measures | Day 1
  Attitudes and stress from dental surgeons will be measured via questionnaire

SECONDARY OUTCOMES:
Sociodemographic characteristics | Day 1
  Age, gender, qualification, personal work status, ethnicity and life characteristics will be assessed by questionnaires
occupation perception | Day 1
  the perception about occupation will be assessed by questionnaires
work conditions | Day 1
  work conditions will be assessed by questionnaires
Changes in practices | Day 1
  changes in practices related to coronavirus pandemic will be assessed by questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Clermont Ferrand, Clermont-Ferrand, France